CLINICAL TRIAL: NCT01595828
Title: An Open Label Study of the Chronic and Acute Effects of Pitavastatin on Monocyte Phenotype, Endothelial Dysfunction and HDL Atheroprotective Function in Subjects With Metabolic Syndrome (CAPITAIN)
Brief Title: Effects of Pitavastatin on Monocyte, Endothelial Dysfunction and HDL-C in Subjects With Metabolic Syndrome
Acronym: CAPITAIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-104-4.03EU
Record Dates: First submitted 2012-05-02; First posted 2012-05-10 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pitavastatin 4mg daily (Experimental): 4 mg tablets of pitavastatin by oral route for a period of 6 months
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin

SUMMARY:
The purpose of this study is to examine in detail the acute and chronic effects of pitavastatin on plasma lipid transport and atheroma biomarkers in patients at elevated risk for the premature development of atherosclerosis (CAPITAIN).

ELIGIBILITY:
Inclusion Criteria:

* Patients with metabolic syndrome
* Patients with LDL-C > 130mg/dL
* Eligible, able to participate and have given informed consent

Exclusion Criteria:

* Body Mass Index >35 kg/m2
* LDL-C > 190mg/dL
* Fasting triglycerides > 400 mg/dL
* Diabetes mellitus (fasting glucose >7 mmol/L) or taking diabetic therapy
* Uncontrolled hypertension (Systolic Blood Pressure >= 140 mmHg or Diastolic Blood Pressure >= 90mmHg)
* Any conditions that cause secondary dyslipidaemia or increase the risk of statin therapy
* ALAT and ASAT >3 x ULRR
* Impaired renal function (Serum Creatinine >1.5 x ULRR or eGFR <60 mL/min)
* History of any muscle disease or unexplained elevation (>3 x ULRR) of serum creatine kinase
* Evidence of symptomatic heart failure (NYHA class III or IV)
* Current or recent user of supplements or medications known to alter lipid metabolism

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 180 in plasma biomarkers of inflammation and atherosclerosis, including monocytes, lymphocytes, endothelial adhesion proteins, atherogenic lipoproteins and cardioprotective HDL | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Kowa Research Europe Ltd., Wokingham, United Kingdom

REFERENCES:
- [Derived] Chapman MJ, Orsoni A, Mellett NA, Nguyen A, Robillard P, Shaw JE, Giral P, Therond P, Swertfeger D, Davidson WS, Meikle PJ. Pitavastatin treatment remodels the HDL subclass lipidome and proteome in hypertriglyceridemia. J Lipid Res. 2024 Feb;65(2):100494. doi: 10.1016/j.jlr.2023.100494. Epub 2023 Dec 29. PMID 38160756
- [Derived] Therond P, Chapman MJ. Sphingosine-1-phosphate: metabolism, transport, atheroprotection and effect of statin treatment. Curr Opin Lipidol. 2022 Jun 1;33(3):199-207. doi: 10.1097/MOL.0000000000000825. Epub 2022 Mar 9. PMID 35695616
- [Derived] Chapman MJ, Orsoni A, Tan R, Mellett NA, Nguyen A, Robillard P, Giral P, Therond P, Meikle PJ. LDL subclass lipidomics in atherogenic dyslipidemia: effect of statin therapy on bioactive lipids and dense LDL. J Lipid Res. 2020 Jun;61(6):911-932. doi: 10.1194/jlr.P119000543. Epub 2020 Apr 15. PMID 32295829
- [Derived] Chapman MJ, Orsoni A, Robillard P, Therond P, Giral P. Duality of statin action on lipoprotein subpopulations in the mixed dyslipidemia of metabolic syndrome: Quantity vs quality over time and implication of CETP. J Clin Lipidol. 2018 May-Jun;12(3):784-800.e4. doi: 10.1016/j.jacl.2018.02.001. Epub 2018 Feb 9. PMID 29574070
- [Derived] Orsoni A, Therond P, Tan R, Giral P, Robillard P, Kontush A, Meikle PJ, Chapman MJ. Statin action enriches HDL3 in polyunsaturated phospholipids and plasmalogens and reduces LDL-derived phospholipid hydroperoxides in atherogenic mixed dyslipidemia. J Lipid Res. 2016 Nov;57(11):2073-2087. doi: 10.1194/jlr.P068585. Epub 2016 Aug 31. PMID 27581680
- [Derived] Meikle PJ, Wong G, Tan R, Giral P, Robillard P, Orsoni A, Hounslow N, Magliano DJ, Shaw JE, Curran JE, Blangero J, Kingwell BA, Chapman MJ. Statin action favors normalization of the plasma lipidome in the atherogenic mixed dyslipidemia of MetS: potential relevance to statin-associated dysglycemia. J Lipid Res. 2015 Dec;56(12):2381-92. doi: 10.1194/jlr.P061143. Epub 2015 Oct 20. PMID 26486974
- [Derived] Chapman MJ, Orsoni A, Robillard P, Hounslow N, Sponseller CA, Giral P. Effect of high-dose pitavastatin on glucose homeostasis in patients at elevated risk of new-onset diabetes: insights from the CAPITAIN and PREVAIL-US studies. Curr Med Res Opin. 2014 May;30(5):775-84. doi: 10.1185/03007995.2013.874989. Epub 2014 Jan 10. PMID 24328357